CLINICAL TRIAL: NCT06019767
Title: Peer-led Trauma Therapy for Re-entry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1144; Protocol Version 12/02/24 (Other: UW Madison); SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison)
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: PTSD
Keywords: Previously incarcerated; Group therapy; Cognitive Processing Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Processing Therapy (CPT) (Experimental): Groups of 6-8 receive CPT to treat PTSD
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — CPT is a type of cognitive behavioral therapy recommended for the treatment of PTSD. Delivered over 12 sessions with an emphasis on addressing trauma-related cognitions and challenging trauma-related beliefs. Includes homework assignments. For this study, CPT will be conducted in groups.

SUMMARY:
The purpose of the research is to learn more about how to treat PTSD for people directly impacted by incarceration (i.e., have spent time in prison or jail). This research will help identify if a PTSD treatment group that is used in community settings, and led by individuals with lived experience, is helpful in reducing PTSD symptoms among people who have been directly impacted by incarceration.

Participants will complete an interview to determine whether they are experiencing PTSD, and if so, will participate in a 6-week therapy group treatment.

DETAILED DESCRIPTION:
Two community Certified Peer Specialists (CPSs) who have experienced incarceration and re-entry from prison, and who have experienced trauma will be trained on delivering group Cognitive Processing Therapy (CPT).

Working with the Wisconsin Department of Health Services (DHS) and community organizations serving formerly incarcerated individuals, researchers will screen individuals for PTSD treatment need, and invite 48 eligible individuals to participate in group CPT co-led by one of the trained CPSs and a trained community therapist or provider.

Eligible participants who are enrolled in the study will be invited to complete a 6-week (12 sessions total) group CPT therapy treatment for PTSD. Participants will also complete pre-, mid-, and post-treatment mental health surveys. Participants will also complete a post-treatment focus group or post-treatment individual interview where they are asked about their experience in the therapy and to provide feedback on the study as a whole.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* completed a prison or jail sentence
* no current psychosis symptoms
* no active self-harm or active suicidal intent
* able and willing to participate in group therapy
* meet criteria for PTSD treatment need

Exclusion Criteria:

* current and active psychosis
* current and active self-harm and suicidality
* no PTSD diagnosis
* current substance use dependence (not including those used as prescribed for medical reasons) on alcohol, cocaine, amphetamines, inhalants, sedatives or sleeping pills, hallucinogens, or opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Feasibility: Participation | Study duration (up to 2 years)
  Will be measured as the percentage of invited, eligible individuals who elect to participate.
Feasibility: Rate of retention | Study duration (up to 2 years)
  Will be measured by percentage of participants who complete at least 9 of the 12 study sessions
Feasibility: Compliance through participation | Study duration (up to 2 years)
  Will be measured by percentage of participants performing intervention activities during session, such as contributing to the discussion.
Feasibility: Compliance through homework | Study duration (up to 2 years)
  Will be measured by percentage of participants completing homework assignments each week.
Feasibility: Compliance through completing assessments | Study duration (up to 2 years)
  Will be measured by percentage of participants completing the pre-, mid-, and post-intervention assessment batteries.
Ratings from 0-5 by clinical supervisors on therapist adherence to five session elements | Study duration (up to 2 years)
  Higher ratings indicate better adherence to session elements. Assesses for therapist adherence to CPT guidelines as secondary measure of intervention efficacy.
Ratings 1-7 by clinical supervisors on quality of session elements delivered by therapist | Study duration (up to 2 years)
  Higher ratings indicate higher-quality session element (scores 1-7; 1=not satisfactory, 4= satisfactory, 7=excellent) by the clinical supervisor. Assesses for therapist compliance as secondary measure of intervention efficacy.
Change in suicide and self-harm ideation | Baseline to end of follow-up (up to 4.5 months)
  Beck Depression Inventory-II (BDI-II), item 9. Participants will answer the item on a scale of 0-3, where a score of 2 or 3 indicates higher ideation.
Participant satisfaction | One week post-treatment (up to 7 weeks)
  Using the 8 item Client Satisfaction Questionnaire (CSQ-8), participants will rate their satisfaction with their experience. Scale ranges from 1-4, with total potential scores of 8 to 32 with higher scores indicating greater satisfaction.
Change in PTSD symptom severity | Baseline to end of follow-up (up to 4.5 months)
  Using the PTSD Checklist for DSM-5 (PCL-5), which is a 20-item self-report measure, symptoms of PTSD will be assessed. Participants will answer items on a scale of 0-4, where 0=Not at all and 4=Extremely. Higher scores indicate higher symptom severity.

SECONDARY OUTCOMES:
Change in depression symptom severity | Baseline to end of follow-up (up to 4.5 months)
  Beck Depression Inventory-II (BDI-II), which is a 21-item self-report measure to assess depression severity. Participants will answer items on a scale of 0-3, where lower scores indicate lower severity.
Change in trauma related thoughts and beliefs | Baseline to end of follow-up (up to 4.5 months)
  Posttraumatic Cognitions Inventory (PTCI) is a 33-item measure of negative cognition about the world, negative self-related thoughts, and self-blame. Participants rate each item on a scale of 1-7, 1=totally disagree, 4=neutral, 7=totally agree. Higher scores indicate greater levels of trauma.
Change in aspects of hopelessness | Baseline to end of follow-up (up to 4.5 months)
  Beck Hopelessness Scale is a 20-item questionnaire, which participants answer true or false.
Change in substance use | Baseline to end of follow-up (up to 4.5 months)
  Tobacco, Alcohol, Prescription Medication, and other Substance Use Tool (TAPS) screens for tobacco use, alcohol use, prescription medication misuse, and illicit substance use in the past year, as well as the past 3 months.
Change in anxiety symptom severity | Baseline to end of follow-up (up to 4.5 months)
  Beck Anxiety Inventory (BAI), which is a 21-item self-report measure to assess anxiety severity. Participants will rate how much items bothered them as: Not at all; Mildly but it didn't bother me much; Moderately - it wasn't pleasant at times; or, Severely - it bothered me a lot. More symptoms that caused moderate or severe bother indicate higher severity of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koenigs, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No